CLINICAL TRIAL: NCT03912532
Title: A Phase 2b, Randomized, Double-blind, Placebo-controlled, Multi-center Study to Evaluate the Efficacy, Safety, and Tolerability of Three Doses of NGM282 Administered for 24 Weeks for the Treatment of Histologically Confirmed Nonalcoholic Steatohepatitis (NASH)
Brief Title: Evaluation of Efficacy, Safety and Tolerability of Aldafermin in a Phase 2b, Randomized, Double-blind, Placebo-controlled, Multi-center Study In Subjects With Nonalcoholic Steatohepatitis and Stage 2/3 Fibrosis (ALPINE 2/3)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NGM Biopharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18-0108
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Results first posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-03

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — aldafermin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- NGM282 Dose 1 (Experimental): Administered by subcutaneous injection
  Interventions: Biological: NGM282
- NGM282 Dose 2 (Experimental): Administered by subcutaneous injection
  Interventions: Biological: NGM282
- NGM282 Dose 3 (Experimental): Administered by subcutaneous injection
  Interventions: Biological: NGM282
- Placebo (Placebo Comparator): Administered by subcutaneous injection
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: NGM282 — NGM282
  Arms: NGM282 Dose 1; NGM282 Dose 2; NGM282 Dose 3
Other: Placebo — Placebo for NGM282
  Arms: Placebo

SUMMARY:
This is a multi-center evaluation of NGM282 in a randomized, double-blind, placebo-controlled study administered for 24 weeks in participants with histologically confirmed NASH and F2/F3 Fibrosis.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed NASH diagnosis as defined by the NASH CRN
2. Total liver fat content of ≥ 8% as measured by MRI-PDFF

Exclusion Criteria:

1. Clinically significant acute or chronic liver disease of an etiology other than NASH
2. Evidence of drug-induced steatohepatitis secondary to amiodarone, corticosteroids, estrogens, methotrexate, tetracycline, or other medications known to cause hepatic steatosis
3. History or presence of cirrhosis (compensated or decompensated) as determined by histology and/or relevant medical complications and/or laboratory parameters
4. Prior or pending liver transplantation

Other protocol-defined inclusion/exclusion criteria could apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2021-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: NGM Study Director, Study Director — NGM Biopharmaceuticals
Locations (34):
- United States (33):
  - NGM Clinical Study Site, Chandler, Arizona
  - NGM Clinical Study Site 814, Tucson, Arizona
  - NGM Clinical Study Site 816, Tucson, Arizona
  - NGM Clinical Study Site, North Little Rock, Arkansas
  - NGM Clinical Study Site, Fresno, California
  - NGM Clinical Study Site, La Jolla, California
  - NGM Clinical Study Site, Los Angeles, California
  - NGM Clinical Study Site, Poway, California
  - NGM Clinical Study Site, Rialto, California
  - NGM Clinical Study Site, Boca Raton, Florida
  - NGM Clinical Study Site, Lakewood Rch, Florida
  - NGM Clinical Study Site, Port Orange, Florida
  - NGM Clinical Study Site, Sarasota, Florida
  - NGM Clinical Study Site, The Villages, Florida
  - NGM Clinical Study Site, Chicago, Illinois
  - NGM Clinical Study Site, Baton Rouge, Louisiana
  - NGM Clinical Study Site, Baltimore, Maryland
  - NGM Clinical Study Site, Ann Arbor, Michigan
  - NGM Clinical Study Site, Flowood, Mississippi
  - NGM Clinical Study Site, Jackson, Mississippi
  - NGM Clinical Study Site, Kansas City, Missouri
  - NGM Clinical Study Site, St Louis, Missouri
  - NGM Clinical Study Site, New York, New York
  - NGM Clinical Study Site, Durham, North Carolina
  - NGM Clinical Study Site, Fayetteville, North Carolina
  - NGM Clinical Study Site, Germantown, Tennessee
  - NGM Clinical Study Site, Hermitage, Tennessee
  - NGM Clinical Study Site, Austin, Texas
  - NGM Clinical Study Site 845, Edinburg, Texas
  - NGM Clinical Study Site, Edinburg, Texas
  - NGM Clinical Study Site, Houston, Texas
  - NGM Clinical Study Site, San Antonio, Texas
  - NGM Clinical Study Site, Richmond, Virginia
- NGM Clinical Study Site, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Harrison SA, Abdelmalek MF, Neff G, Gunn N, Guy CD, Alkhouri N, Bashir MR, Freilich B, Kohli A, Khazanchi A, Sheikh MY, Leibowitz M, Rinella ME, Siddiqui MS, Kipnes M, Moussa SE, Younes ZH, Bansal M, Baum SJ, Borg B, Ruane PJ, Thuluvath PJ, Gottwald M, Khan M, Chen C, Melchor-Khan L, Chang W, DePaoli AM, Ling L, Lieu HD. Aldafermin in patients with non-alcoholic steatohepatitis (ALPINE 2/3): a randomised, double-blind, placebo-controlled, phase 2b trial. Lancet Gastroenterol Hepatol. 2022 Jul;7(7):603-616. doi: 10.1016/S2468-1253(22)00017-6. Epub 2022 Mar 21. PMID 35325622

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 171 participants who met all inclusion criteria and no exclusion criteria were randomized to receive treatment at 37 clinic sites in the United States.
Groups:
- Aldafermin 0.3 mg: Participants who were randomized to receive a single subcutaneous injection of aldafermin 0.3 mg.
- Aldafermin 1.0 mg: Participants who were randomized to receive a single subcutaneous injection of aldafermin 1.0 mg.
- Aldafermin 3.0 mg: Participants who were randomized to receive a single subcutaneous injection of aldafermin 3.0 mg.
- Placebo: Participants who were randomized to receive a single subcutaneous injection of placebo.
Period: Overall Study
Arm/Group | Aldafermin 0.3 mg | Aldafermin 1.0 mg | Aldafermin 3.0 mg | Placebo
Started | 43 | 42 | 43 | 43
Completed | 35 | 35 | 37 | 36
Not Completed | 8 | 7 | 6 | 7
Not completed — Adverse Event | 3 | 3 | 2 | 2
Not completed — Lost to Follow-up | 3 | 2 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 2 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 3
Not completed — Other | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were assessed in the Intent-to-Treat Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Aldafermin 0.3 mg | Aldafermin 1.0 mg | Aldafermin 3.0 mg | Placebo | Total
Number analyzed (Participants) | 43 | 42 | 43 | 43 | 171
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 0 | 0 | 1
  Between 18 and 65 years | 34 | 35 | 36 | 35 | 140
  >=65 years | 9 | 6 | 7 | 8 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (11.2) | 49.8 (13.2) | 52.7 (11.1) | 53.0 (10.8) | 52.5 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 29 | 29 | 26 | 112
  Male | 15 | 13 | 14 | 17 | 59
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 40 | 38 | 39 | 41 | 158
  Black or African American | 0 | 2 | 0 | 2 | 4
  Asian | 0 | 0 | 1 | 0 | 1
  American Indian or Alaska Native | 1 | 0 | 2 | 0 | 3
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Other | 2 | 2 | 1 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Liver Fibrosis Response After Administration With Aldafermin in Participants With Nonalcoholic Steatohepatitis and Stage 2/3 Fibrosis
Description: Liver biopsies were collected at baseline and Week 24 and read by a central pathologist using Nonalcoholic Steatohepatitis Clinical Research Network (NASH CRN) criteria. Fibrosis stages of F0, F1, F2, F3 and F4 are defined by NASH CRN criteria with F0 (minimal score) indicating no fibrosis and F4 (maximal score) indicating liver cirrhosis. Liver fibrosis response was defined as an improvement in liver fibrosis >=1 stage with no worsening of steatohepatitis on liver biopsy at Week 24 compared with baseline.
Time Frame: Baseline up to Week 24
Population: Liver fibrosis response was assessed in the Intent-to-Treat Analysis Set.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Aldafermin 0.3 mg | Aldafermin 1.0 mg | Aldafermin 3.0 mg | Placebo
Number analyzed (Participants) | 43 | 42 | 43 | 43
score on a scale | 0.24 (0.04) | 0.25 (0.04) | 0.27 (0.07) | 0.23 (0.06)
Statistical Analysis 1: Comparison: Aldafermin 0.3 mg vs Aldafermin 1.0 mg vs Aldafermin 3.0 mg vs Placebo; Test type: Other — The Multiple Comparison Procedure-Modelling (MCP-Mod) is a 2-stage procedure in which dose-response models are selected at the design stage. These candidate models are used for both dose-response testing (MCP step) and estimation (Mod step). The dose-response testing is performed using a multiple comparison method to account for the multiplicity issue associated with the multiple candidate models. Missing responses were imputed using multiple imputation under the assumption of missing at random; p = 0.5534, Multiple comparison procedure step

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events After Administration With Aldafermin in Participants With Nonalcoholic Steatohepatitis and Stage 2/3 Fibrosis
Description: Treatment-emergent adverse events (TEAEs) were defined as adverse events (AEs) that commenced on or after the date and time of first study drug administration.
Time Frame: Baseline up to Week 24
Population: TEAEs were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Aldafermin 0.3 mg | Aldafermin 1.0 mg | Aldafermin 3.0 mg | Placebo
Number analyzed (Participants) | 43 | 41 | 43 | 43
Participants
  Any TEAE | 30 | 34 | 38 | 36
  Any TEAE, Grade 1 | 11 | 12 | 17 | 10
  Any TEAE, Grade 2 | 16 | 18 | 19 | 24
  Any TEAE, Grade 3 | 1 | 2 | 2 | 1
  Any TEAE, Grade 4 | 2 | 1 | 0 | 1
  Any TEAE, Grade 5 | 0 | 1 | 0 | 0
  Any aldafermin-related TEAE | 13 | 20 | 21 | 14
  Any TEAE, not related to aldafermin | 17 | 14 | 17 | 22
  Any TEAE, possible related to aldafermin | 10 | 8 | 7 | 11
  Any TEAE, probable related to aldafermin | 2 | 5 | 5 | 2
  Any TEAE, definite related to aldafermin | 1 | 7 | 9 | 1
  Any rosuvastatin-related TEAE | 13 | 4 | 9 | 8
  Any TEAE, not related to rosuvastatin | 17 | 30 | 29 | 28
  Any TEAE, possible related to rosuvastatin | 10 | 1 | 6 | 6
  Any TEAE, probable related to rosuvastatin | 1 | 1 | 3 | 1
  Any TEAE, definite related to rosuvastatin | 2 | 2 | 0 | 1
  Any TEAE leading to study drug withdrawal | 3 | 4 | 3 | 3
  Any aldafermin-related TEAE leading to study drug withdrawal | 1 | 1 | 1 | 2
  Any rosuvastatin-related TEAE leading to study drug withdrawal | 2 | 0 | 0 | 1
  Any serious TEAE | 1 | 4 | 1 | 3
  Any TEAEs leading to death | 0 | 1 | 0 | 0

3. Secondary Outcome: Mean Percentage of Liver Fat Content in Participants With Nonalcoholic Steatohepatitis and Stage 2/3 Fibrosis
Description: Mean percentage of liver fat content was assessed by magnetic resonance imaging-proton density fat fraction (MRI-PDFF).
Time Frame: Baseline, Week 12, Week 24, and Week 30
Population: Mean change in liver fat content was assessed in the Intent-to-Treat Analysis Set.
Measure: Mean (Standard Deviation); unit: percentage of liver fat content
Arm/Group | Aldafermin 0.3 mg | Aldafermin 1.0 mg | Aldafermin 3.0 mg | Placebo
Number analyzed (Participants) | 43 | 42 | 43 | 43
percentage of liver fat content
  Baseline | 19.13 (7.6) | 17.40 (6.4) | 18.69 (7.5) | 17.00 (6.6)
  Week 12: number analyzed (Participants) | 38 | 37 | 37 | 39
  Week 12 | 14.43 (8.8) | 10.62 (5.6) | 7.03 (5.7) | 16.00 (7.1)
  Week 24: number analyzed (Participants) | 37 | 33 | 37 | 37
  Week 24 | 14.85 (9.3) | 10.64 (6.2) | 6.72 (5.6) | 14.01 (6.2)
  Week 30: number analyzed (Participants) | 34 | 31 | 36 | 36
  Week 30 | 16.30 (9.2) | 15.36 (6.5) | 13.10 (7.4) | 14.27 (7.5)

4. Secondary Outcome: Change From Baseline in Liver Fat Content in Participants With Nonalcoholic Steatohepatitis and Stage 2/3 Fibrosis
Description: Change from baseline in liver fat content was assessed by magnetic resonance imaging-proton density fat fraction (MRI-PDFF). Negative values indicate an improvement in liver fat content.
Time Frame: Baseline to Week 12, Week 24, and Week 30
Population: Mean change from baseline in liver fat content was assessed in the Intent-to-Treat Analysis Set.
Measure: Mean (Standard Error); unit: percentage of liver fat content
Arm/Group | Aldafermin 0.3 mg | Aldafermin 1.0 mg | Aldafermin 3.0 mg | Placebo
Number analyzed (Participants) | 38 | 37 | 37 | 39
percentage of liver fat content
  Change from baseline to Week 12 | -4.28 (0.83) | -7.50 (0.85) | -11.37 (0.84) | -1.49 (0.82)
  Change from baseline to Week 24: number analyzed (Participants) | 37 | 33 | 37 | 37
  Change from baseline to Week 24 | -3.73 (0.97) | -7.35 (1.04) | -11.37 (0.98) | -3.44 (0.98)
  Mean change from baseline to Week 30: number analyzed (Participants) | 34 | 31 | 36 | 36
  Mean change from baseline to Week 30 | -2.10 (1.08) | -2.95 (1.13) | -5.19 (1.05) | -2.92 (1.05)

5. Secondary Outcome: Number of Participants With Liver Fat Normalization and Response in Participants With Nonalcoholic Steatohepatitis and Stage 2/3 Fibrosis
Description: Liver fat normalization (LFC; defined as <5%) and response (LFC decrease >=5% from baseline and LFC relative decrease >=30% from baseline) were assessed by magnetic resonance imaging-proton density fat fraction (MRI-PDFF). The responders were defined as participants with either normalization (<5%) or response (decrease from baseline >=5% or relative decrease from baseline >=30%).
Time Frame: Baseline to Week 12, Week 24 and Week 30
Population: Liver fat content normalization and response were assessed in participants with available data in the Intent-to-Treat Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Aldafermin 0.3 mg | Aldafermin 1.0 mg | Aldafermin 3.0 mg | Placebo
Number analyzed (Participants) | 38 | 37 | 37 | 39
Participants
  Week 12: Normalization, response | 3 | 4 | 17 | 0
  Week 12: Normalization, No response | 35 | 33 | 20 | 39
  Week 12: Decrease >=5%, Response | 19 | 24 | 33 | 7
  Week 12: Decrease >=5%, No response | 19 | 13 | 4 | 32
  Week 12: Relative decrease >=30%, Response | 19 | 25 | 33 | 7
  Week 12: Relative decrease >=30%, No response | 19 | 12 | 4 | 32
  Week 24: Normalization, response: number analyzed (Participants) | 37 | 33 | 37 | 37
  Week 24: Normalization, response | 4 | 4 | 20 | 2
  Week 24: Normalization, No response: number analyzed (Participants) | 37 | 33 | 37 | 37
  Week 24: Normalization, No response | 33 | 29 | 17 | 35
  Week 24: Decrease >=5%, Response: number analyzed (Participants) | 37 | 33 | 37 | 37
  Week 24: Decrease >=5%, Response | 21 | 21 | 30 | 10
  Week 24: Decrease >=5%, No response: number analyzed (Participants) | 37 | 33 | 37 | 37
  Week 24: Decrease >=5%, No response | 16 | 12 | 7 | 27
  Week 24: Relative decrease >=30%, Response: number analyzed (Participants) | 37 | 33 | 37 | 37
  Week 24: Relative decrease >=30%, Response | 18 | 20 | 32 | 11
  Week 24: Relative decrease >=30%, No response: number analyzed (Participants) | 37 | 33 | 37 | 37
  Week 24: Relative decrease >=30%, No response | 19 | 13 | 5 | 26
  Week 30: Normalization, response: number analyzed (Participants) | 34 | 31 | 36 | 36
  Week 30: Normalization, response | 4 | 1 | 4 | 4
  Week 30: Normalization, No response: number analyzed (Participants) | 34 | 31 | 36 | 36
  Week 30: Normalization, No response | 30 | 30 | 32 | 32
  Week 30: Decrease >=5%, Response: number analyzed (Participants) | 34 | 31 | 36 | 36
  Week 30: Decrease >=5%, Response | 8 | 12 | 15 | 9
  Week 30: Decrease >=5%, No response: number analyzed (Participants) | 34 | 31 | 36 | 36
  Week 30: Decrease >=5%, No response | 26 | 19 | 21 | 27
  Week 30: Relative decrease >=30%, Response: number analyzed (Participants) | 34 | 31 | 36 | 36
  Week 30: Relative decrease >=30%, Response | 10 | 11 | 16 | 10
  Week 30: Relative decrease >=30%, No response: number analyzed (Participants) | 34 | 31 | 36 | 36
  Week 30: Relative decrease >=30%, No response | 24 | 20 | 20 | 26

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from screening up to Week 30.
Description: TEAEs defined as AEs that started on or after the date of first study drug dosing. AEs without an onset date were defined as TE, except if an incomplete date (eg, mon/yr) clearly indicated the event started prior to the start of first dose of study drug or if the AE stop date indicated that the event started or stopped prior to the start of first dose of study drug.
  The at Risk in the Aldafermin 1.0 mg group is 41 from the Safety Analysis Set, and the Intent-to-Treat group is 42.
Arm/Group | Aldafermin 0.3 mg | Aldafermin 1.0 mg | Aldafermin 3.0 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/43 | 1/41 | 0/43 | 0/43
Serious Adverse Events (participants affected / at risk) | 1/43 | 4/41 | 1/43 | 3/43
Other Adverse Events (participants affected / at risk) | 30/43 | 34/41 | 38/43 | 36/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aldafermin 0.3 mg (N=43) | Aldafermin 1.0 mg (N=41) | Aldafermin 3.0 mg (N=43) | Placebo (N=43)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0 | 0
Cardiac hypertrophy (Cardiac disorders) | 0 | 1 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1
Bronchogenic cyst (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aldafermin 0.3 mg (N=43) | Aldafermin 1.0 mg (N=41) | Aldafermin 3.0 mg (N=43) | Placebo (N=43)
Abdominal distension (Gastrointestinal disorders) | 2 | 2 | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 3 | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 5 | 3 | 2 | 4
Constipation (Gastrointestinal disorders) | 5 | 1 | 1 | 2
Diarrhea (Gastrointestinal disorders) | 3 | 5 | 10 | 6
Flatulence (Gastrointestinal disorders) | 1 | 0 | 3 | 0
Frequent bowel movements (Gastrointestinal disorders) | 1 | 1 | 4 | 0
Nausea (Gastrointestinal disorders) | 5 | 8 | 7 | 8
Vomiting (Gastrointestinal disorders) | 3 | 0 | 1 | 2
Fatigue (General disorders) | 3 | 0 | 4 | 4
Influenza-like illness (General disorders) | 0 | 0 | 3 | 0
Injection site bruising (General disorders) | 1 | 2 | 3 | 2
Injection site erythema (General disorders) | 0 | 4 | 6 | 0
Injection site pruritus (General disorders) | 0 | 2 | 3 | 0
Influenza (Infections and infestations) | 3 | 2 | 1 | 1
Nasopharyngitis (Infections and infestations) | 4 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 5 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 3
Urinary tract infection (Infections and infestations) | 1 | 1 | 2 | 4
Procedural pain (Injury, poisoning and procedural complications) | 0 | 2 | 2 | 4
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 3 | 2 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1 | 2
Headache (Nervous system disorders) | 6 | 2 | 4 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2 | 1
Hypertension (Vascular disorders) | 0 | 3 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-01-15): https://cdn.clinicaltrials.gov/large-docs/32/NCT03912532/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/32/NCT03912532/SAP_001.pdf